CLINICAL TRIAL: NCT02467478
Title: Role of Linagliptin in Improving Renal Failure by Improving CD34+ Stem Cell Number, Function and Gene Expression in Renal Function Impaired Type 2 Diabetes Patients.
Brief Title: Linagliptin's Effect on CD34+ Stem Cells
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Sabyasachi Sen, Associate Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 121439
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes; Impaired Renal Function
Keywords: Diabetes Mellitus, Type 2; Endothelial cells; Cellular biomarker; endothelial dysfunction; CD34+; Impaired renal function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo 1 pill daily for 12 weeks
  Interventions: Drug: Placebo
- Linagliptin (Active Comparator): Linagliptin 5mg once daily for 12 weeks
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — 5 mg tablet once daily for 12 weeks
  Other Names: TRADJENTA
  Arms: Linagliptin
Drug: Placebo — 1 tablet daily for 12 weeks
  Arms: Placebo

SUMMARY:
Type 2 diabetes is a national epidemic. Diabetes has undesirable effects on blood vessels which may contribute to heart disease. Endothelial Progenitor Cells (EPCs) are found in the blood. Research has shown that improving the survival of these special blood cells may decrease the harmful effects of diabetes on blood vessels and reduce or reverse heart disease. Linagliptin is an Food and Drug Administration (FDA) approved prescription medicine used along with insulin or with oral medications to lower blood sugar in people with Type 2 diabetes. It is in a class of diabetes medication called Dipeptidyl peptidase-4 (DPP-4) inhibitors. DPP-4 inhibitors have been shown to increase EPCs in patients with Type 2 diabetes.

Hypothesis: Both type 2 diabetes and Chronic Kidney Disease (CKD) are associated with poor stem cell number and function. Poor viability and function of EPCs in CKD and diabetes The investigators hypothesize that use of Linagliptin (along with Insulin) may help reduce cardiovascular risk by improving EPC survival and function above and beyond adequate glucose metabolism control

DETAILED DESCRIPTION:
Type 2 diabetes is a national epidemic with significant macro and microvascular complications. Insulin resistance in pre-diabetes and overt diabetes are associated with endothelial dysfunction.

A few studies indicate that stem cells particularly EPCs can act as a suitable bio-marker for monitoring cardiovascular morbidity. In this proposal the investigators suggest that EPCs or CD34 positive cells (defined as CD34/vascular endothelial growth factor receptor 2 (VEGFR2+) cells) can act as a suitable cellular biomarker for estimating and following endothelial dysfunction in early type 2 diabetes patients with CKD. EPCs have been shown to be dysfunctional in both CKD patients and type 2 Diabetes Mellitus (DM) patients.

Linagliptin (TRADJENTA) tablets are indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus. No dose adjustment is recommended for patients with renal impairment.

EPCs have been used as a regenerative tool in ischemic myocardium and diabetic wound healing. Endothelial dysfunction with associated inflammation may be a consequence of excess intra-cellular super-oxide presence in a setting of diabetes which is a pro-oxidative stress condition ultimately leading to poor EPC function and senescence.

Though lifestyle modification has been proposed as a main stay for prevention and treatment of early type 2 diabetes, several new therapies for diabetes have been developed in recent years. Incretins and incretin mimetics appear to hold promise. Mechanism of positive effect of exercise and oral hypoglycemic agents can be very different.

DPP-4 inhibitors have been shown to increase EPCs in patients with type 2 diabetes reportedly via stromal cell-derived factor 1 (SDF-1) alpha up-regulation. Interestingly, up-regulation of SDF-1 alpha and vascular endothelial growth factor (VEGF), both chemotactic factors increase mobilization and recruitment of EPCs in the face of acute ischemic injury for repair and regeneration.

Several studies have shown positive effect of incretins (Glucagon like peptide, GLP-1) and incretin receptor agonists (GLP-1 receptor agonists) on cardiovascular risk factors in type 2 diabetes patients and even in patients with chronic heart failure and left ventricular dysfunction who do not have diabetes.

DPP-4 Inhibitors may have cardio-protective effects of their own, as they increase bio-availability of endogenous GLP-1. They improve blood flow and nitric oxide production in endothelium. These are unique properties not demonstrated by other oral diabetes medications. The mechanism underlying these effects may be mediated by increased nitric oxide bioavailability but is not completely known. However these beneficial effects appear to be independent of glycemia reduction.

It is however unknown whether Linagliptin will have any positive effect on human EPC function where two prominent cardiovascular risk factors co-exist such as CKD and type 2 diabetes.

Therefore the investigators plan to investigate if Linagliptin can alter function and gene expression of CD34+ cells in a setting of CKD and type 2 diabetes. The investigators choose to look at non geriatric adult population with early type 2 diabetes (less than 10 years of duration) at an early phase of renal impairment (stages 1-3).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-70 years
* Diagnosis of type 2 diabetes within the previous 15 years using criteria of the American Diabetes Association
* Currently being treated with 1-2 grams/day of metformin, or insulin or both stably
* Hemoglobin A1c (HbA1C) between 6.5% to 10.0% (both inclusive)
* Body Mass Index (BMI) between 25 and 39.9 kg/m2 (both inclusive)
* Chronic Kidney disease (CKD) Stages 1-3, Creatinine clearance (CrCl) less than 90 and more than 29

Exclusion Criteria:

* Type 1 diabetes
* History of Diabetic Ketoacidosis (DKA) or hyperosmolar nonketotic coma
* Hemoglobinopathies with low hematocrit (Below 28 Units)
* History of pancreatitis
* History of cancer within the past 5 years (except basal cell carcinoma)
* Previous cardiovascular or cerebrovascular event within 6 months of screening or active or clinically significant coronary and/or Peripheral Vascular Disease (PVD)
* Statin use started in the last 3 month
* Current use of oral or injectable anti-diabetic medication other than Metformin and insulin
* Consistent use of steroids within the last 3 months
* Any active wounds, or surgery within the past 3 months
* Inflammatory disease, or the chronic use of anti-inflammatory drugs within the past 3 months
* Untreated hyper/hypothyroidism
* Contraindications to moderate exercise
* Implanted devices that might interact with the tanita scale
* Pre-existing liver disease and/or Alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) > 2.5 times Under the Normal Limits (UNL)
* Untreated Systolic blood pressure > 140 mmHg or diastolic blood pressure> 90 mmHg
* Serum creatinine levels ≥ 2.0
* CKD Stages 4 and 5 (estimated CrCl <30 mL/min)
* Triglycerides > 450 mg/dL
* Known allergies or hypersensitivities to Linagliptin or Dipeptidyl peptidase-4 (DDP-4) inhibitors
* Treatment with cytochrome p450 (CYP 3A4) inhibitors
* Women of child bearing age who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study
* Prisoners or subjects that are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Additionally, patients who are active smokers, patients who are pregnant, nursing women, and post-menopausal women who are on hormone replacement therapy will be excluded.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, PhD, Principal Investigator — Medical Faculty Associates
Locations (1):
- The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers.

REFERENCES:
- [Derived] Awal HB, Nandula SR, Domingues CC, Dore FJ, Kundu N, Brichacek B, Fakhri M, Elzarki A, Ahmadi N, Safai S, Fosso M, Amdur RL, Sen S. Linagliptin, when compared to placebo, improves CD34+ve endothelial progenitor cells in type 2 diabetes subjects with chronic kidney disease taking metformin and/or insulin: a randomized controlled trial. Cardiovasc Diabetol. 2020 Jun 3;19(1):72. doi: 10.1186/s12933-020-01046-z. PMID 32493344

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Linagliptin
Started | 17 | 14
Completed | 17 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Customized [Mean (Standard Deviation); unit: years] | 63 (6) | 61 (5) | 62.09 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] — must be between 25-39.9 to participate in the study
  kg/m^2 | 30.6 (2.9) | 31.2 (4.4) | 30.8 (.42)
HbA1c [Mean (Standard Deviation); unit: percentage of hemoglobin] — Must be between 6.5-10.0% to participate in the study
  percentage of hemoglobin | 7.4 (1) | 7.1 (0.7) | 7.26 (.21)
Required to be on stable dose of Metformin and/or Insulin [Number; unit: participants] — Population: Values vary here as patients could be on either an insulin, metformin, or a combination of the two. As a result, some participants may be included in both analysis categories.
  participants
    Metformin | 14 | 12 | 26
    Insulin | 6 | 4 | 10
BP [Mean (Standard Deviation); unit: mmHg]
  Systolic | 133 (18) | 128 (10) | 131 (14)
  Diastolic | 77 (7) | 81 (7) | 79 (7)
Percent Fat [Mean (Standard Deviation); unit: percentage] | 38 (10) | 30 (10) | 34 (10)
Waist cm [Mean (Standard Deviation); unit: centimeters] | 105 (8) | 107 (17) | 106 (12)
Basal Metabolic Rate [Mean (Standard Deviation); unit: Calories/day] | 1476 (448) | 1868 (293) | 1653 (134)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 130 (44) | 125 (26) | 127.5 (12.72)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.3) | 1.1 (0.4) | 1 (.07)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 84 (19) | 83 (21) | 83.5 (1.41)
Cholesterol [Mean (Standard Deviation); unit: mg] | 168 (53) | 166 (52) | 167 (.70)

OUTCOME MEASURES:

1. Primary Outcome: Cellular Markers
Description: The investigators will use participants' peripheral blood derived CD34+ cells looking at number, function, and gene expression. Post Linagliptin will be compared to pre Linagliptin measurements. Here we report fold changes in protein populations as determined by ELISA.
Time Frame: Week 12 expression as a fold difference to Week 0
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
Fold Change
  PECAM | 1.48 (1.11) | 2.48 (2.80)
  VEGFA | 1.43 (1.2) | 2.4 (2.91)
  SOD3 | 1.13 (0.81) | 1.15 (0.86)
  SOD2 | 1.40 (1.34) | 2.47 (4.27)
  GPX3 | 1.59 (1.40) | 1.36 (1.32)

2. Primary Outcome: Urinary Function Marker in CKD
Description: We measure using microalbumin/creatinine ratio provided from a random spot urine sample.
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
ratio | 51.12 (99.55) | 39.70 (68.92)

3. Secondary Outcome: Serum Endothelial Inflammatory Markers
Description: Serum endothelial inflammatory markers included here: high sensitivity C-reactive protein (hs-CRP)
Time Frame: 12 weeks post Linagliptin or Placebo treatment
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
mg/L | 3.08 (3.41) | 5.17 (6.54)

4. Secondary Outcome: Serum Endothelial Inflammatory Markers
Description: Serum endothelial inflammatory markers included here: Interleukin 6 (IL-6)
Time Frame: 12 weeks post Linagliptin or Placebo treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
pg/mL | 2.18 (1.45) | 5.09 (6.08)

5. Secondary Outcome: Fasting Lipid Profile
Description: Measured through serum biochemistry Lipid Panel
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
mg/dl
  Cholesterol | 171.45 (48.49) | 159.69 (48.53)
  Triglycerides | 127.76 (79.04) | 124.31 (50.67)

6. Secondary Outcome: Glycemic Control
Description: Glycemic control is evaluated by measuring HbA1c levels to gauge changes in blood sugar control over last ~90 days
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
percentage of hemoglobin | 7.27 (0.73) | 6.66 (0.40)

7. Secondary Outcome: Glycemic Control: Fasting Glucose
Description: Glycemic control is evaluated by measuring fasting blood glucose at time of measurement
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
mg/dL | 129.68 (46.78) | 109.93 (16.81)

8. Secondary Outcome: Glycemic Control: Insulin
Description: Glycemic control is evaluated by measuring insulin levels at the time of the visit
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
mIU/L | 20.82 (12.6) | 20.52 (19.7)

9. Secondary Outcome: Adiposity
Description: Measured using the Tanita Body Composition Analyzer scale, measured as percentage body fat.
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
percentage of body fat | 30.6 (2.9) | 31.2 (4.4)

10. Secondary Outcome: Estimation of Creatinine Clearance
Description: Measured via blood biochemistry eGFR, an alternative measurement to spot urine urine microalbumin/creatinine ratio presented above
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
mL/min/1.73m^2 | 84.12 (19.81) | 79.46 (19.9)

11. Secondary Outcome: Pulse Wave Analysis
Description: Vessel health is assessed by looking at Arterial stiffness. Augmentation index (AI) is defined as the ratio of the augmentation pressure to the pulse pressure, times 100, to give a percentage. Augmentation index 75 normalizes this value to an estimate of the AI at a heart rate of 75bpm. We used Vascular Flow and wave measurement equipment, SphygmoCor Central Pressure system from AtCor.
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: Percentage (of pulse pressure)
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
Percentage (of pulse pressure)
  Augmentation Index 75 | 21.37 (11.49) | 22.33 (12)
  Augmentation Index | 24.17 (12.93) | 24.93 (14.37)

12. Secondary Outcome: Pulse Wave Velocity
Description: Vessel health is assessed by looking at Arterial stiffness. Pulse wave velocity (PWV) measures the delay between the pulse registered at the femoral artery from the pulse at the carotid. The difference in distance between these two measurement points from the aortic notch is divided by this delay to give a speed. In stiffer, less healthy vessels, the PWV is increased. We used Vascular Flow and wave measurement equipment, SphygmoCor Central Pressure system from AtCor to perform this calculation.
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
m/s | 10.23 (8.65) | 10.53 (8.58)

13. Secondary Outcome: Resting Metabolic Rate (RMR)
Description: (RMR, similar to Resting Energy expenditure measurement): Evaluation of changes in Basal Metabolic Rate
Time Frame: 12 weeks post beginning Linagliptin or placebo treatment
Measure: Mean (Standard Deviation); unit: Calories/day
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 17 | 14
Calories/day | 1650.07 (428.52) | 1657.6 (445.45)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from signing of informed consent to 30 days post final visit (approximately 16 weeks)
Description: The adverse events that occurred during the duration of the study were isolated incidents, therefore, do not have any relation to the study intervention or medication regiment.
Arm/Group | Placebo | Linagliptin
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Linagliptin (N=14)
Kidney Stone (Renal and urinary disorders) | 1 (1) | 1 (1)
Bacterial Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations may include the relatively short duration of 12-week Linagliptin therapy. Limitations also arise because of the small sample size, and due to the difficulty in obtaining all cellular outcome measures, in some patients, due to low total CD34+ cell numbers. Further studies with a larger population and longer duration may be helpful to further define the mechanisms behind our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT02467478/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02467478/ICF_001.pdf